CLINICAL TRIAL: NCT00825305
Title: A Phase III, Single Center, Randomized, Open-label Study, Comparing PCECV Administered in the Abbreviated Zagreb Regimen (2-1-1) to the Conventional Essen Regimen (1-1-1-1-1) in Healthy Volunteers in China
Brief Title: Safety and Immunogenicity (Non-inferiority) of a Purified Chick Embryo Cell Vaccine Vaccine Administered in Two Different Schedules (Conventional Versus Abbreviated Schedule)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M49P8
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Results first posted 2010-05-19 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Rabies
Keywords: vaccine; prevention; rabies; Rabies disease
MeSH Terms: conditions — Rabies

ARMS (2):
- Zagreb (2-1-1) (Experimental): Rabies PCEC vaccine was applied according Zagreb schedule with 2 vaccinations on day 0, 1 vaccination on day 7 and day 21, respectively
  Interventions: Biological: Abbreviated Zagreb 2-1-1 schedule
- Essen (1-1-1-1-1) (Active Comparator): Rabies PCEC vaccine was applied according Essen schedule, i.e. 1 vaccination on day 0, day 3, day 7, day 14 and day 28, respectively.
  Interventions: Biological: Standard Essen 1-1-1-1-1 schedule

INTERVENTIONS:
Biological: Abbreviated Zagreb 2-1-1 schedule — Subjects received the abbreviated Zagreb 2-1-1 schedule in a safety-lead-in phase.
  Other Names: PCEC Rabies vaccine for human use
  Arms: Zagreb (2-1-1)
Biological: Standard Essen 1-1-1-1-1 schedule — Subjects received the standard Essen regimen.
  Other Names: PCEC Rabies vaccine for human use
  Arms: Essen (1-1-1-1-1)

SUMMARY:
This study investigates the safety and immunogenicity (non-inferiority) of a Purified Chick Embryo Cell Vaccine (PCECV) administered in two different schedules (conventional versus abbreviated schedule) in healthy adults 18 to 50 years of age in China

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18-50 years of age who:
* are in good health at the time of entry into the study as determined by medical history, physical examination and clinical judgment of the investigator;
* volunteer for the simulated post-exposure vaccination courses and blood draws;
* have given a written informed consent; informed consent must be obtained for all the subjects before enrolment in the study;
* are available for all the visits scheduled in the study.

Exclusion Criteria:

* Subjects with the below criteria were excluded:
* pregnancy or unwillingness to practice acceptable contraception during participation in the study;
* a history of rabies immunization;
* a significant acute or chronic infectious disease that may impact the subject's safety and /or immunogenicity in the Investigators opinion at the time of enrolment;
* fever ≥ 38.0°C (axillary) or/and significant acute or chronic infection requiring systemic antibiotic or antiviral therapy within the past 7 days before enrolment;
* treatment with corticosteroids, immunosuppressive or antimalaria drugs during the two month period before enrolment;
* administration of any vaccine within the past 14 days before enrolment;
* known/suspected immunodeficiency, or autoimmune disease, or any immunologic disorder;
* history of allergy to egg protein;
* known hypersensitivity to neomycin, tetracycline, amphotericin-B, or any other vaccine component;
* treatment with parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within the past 3 months;
* mental condition rendering the subject unable to understand the nature, scope and consequences of the study;
* participation in any other investigational trial within the past 3 months before enrolment;
* planned surgery during the study period;
* intention to leave the area of the study site before the end of study period;
* any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objective.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 825 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Jizhou, Hebei, China

REFERENCES:
- [Derived] Ma J, Wang H, Li J, Chang L, Xie Y, Liu Z, Zhao Y, Malerczyk C. A randomized open-labeled study to demonstrate the non-inferiority of purified chick-embryo cell rabies vaccine administered in the Zagreb regimen (2-1-1) compared with the Essen regimen in Chinese adults. Hum Vaccin Immunother. 2014;10(10):2805-12. doi: 10.4161/21645515.2014.972773. PMID 25483635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled in November 2008 at 1 center in China.
Pre-assignment Details: All enrolled subjects were randomized, but one subject in the Zagreb (2-1-1) group was not vaccinated.
Groups:
- Abbreviated Zagreb (2-1-1): Abbreviated Zagreb vaccination schedule with 2 vaccinations at day 0, 1 vaccination at day 7 and 1 vaccination at day 21.
- Conventional Essen(1-1-1-1-1): Conventional Essen schedule with 1 vaccination on day 0, day 3, day 7, day 14 and day 28, respectively.
Period: Overall Study
Arm/Group | Abbreviated Zagreb (2-1-1) | Conventional Essen(1-1-1-1-1)
Started | 550 | 275
Completed | 533 | 252
Not Completed | 17 | 23
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 6 | 12
Not completed — Inappropriate inclusion | 1 | 0
Not completed — Protocol Violation | 9 | 9
Not completed — Can not be classified | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abbreviated Zagreb (2-1-1) | Conventional Essen(1-1-1-1-1) | Total
Number analyzed (Participants) | 549 | 275 | 824
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measures are presented for safety population.
  years | 38.2 (7.14) | 39.33 (6.93) | 38.58 (7.09)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline measures are presented for safety population.
  Participants
    Female | 323 | 154 | 477
    Male | 226 | 121 | 347

OUTCOME MEASURES:

1. Primary Outcome: Rabies Virus Neutralizing Antibody Concentrations on Day 14.
Description: Rabies virus neutralizing antibody concentrations of the abbreviated Zagreb regimen compared with the conventional Essen regimen. Results are presented on log2 scale. For results on original geometric (multiplicative) scale please raise numbers to the basis of 2.
Time Frame: 14 days
Population: Due to the Chinese registration requirements, only a subset of subjects bloodsamples were drawn and immunogenicity was evaluated. The per protocol population of this subset was analyzed.
Measure: Log Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Abbreviated Zagreb (2-1-1) | Conventional Essen(1-1-1-1-1)
Number analyzed (Participants) | 69 | 70
IU/mL | 3.1 [2.73 to 3.47] | 3.3 [2.82 to 3.79]
Statistical Analysis 1: Comparison: Abbreviated Zagreb (2-1-1) vs Conventional Essen(1-1-1-1-1); Test type: Non-Inferiority or Equivalence — The null hypothesis states that the Zagreb schedule is inferior to the Essen schedule in terms of day 14 antibody titers assuming no difference between the two schedules and the equivalence limit of 1.5 titer levels (log2); ANOVA; ratio of log2 mean = -0.2, 95% CI 2-sided [-0.81 to 0.4] — Ratio of log2 mean (Zagreb/Essen) on day 14

2. Secondary Outcome: Rabies Virus Neutralizing Antibody Concentrations on Day 7 and Day 42.
Description: Rabies virus neutralizing antibody concentrations the abbreviated Zagreb regimen compared with the conventional Essen regimen. Results are presented on log2 scale. For results on original geometric (multiplicative) scale please raise numbers to the basis of 2.
Time Frame: 7 days and 42 days
Population: as for outcome 1
Measure: Log Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | Abbreviated Zagreb (2-1-1) | Conventional Essen(1-1-1-1-1)
Number analyzed (Participants) | 69 | 70
IU/ml
  day 7 results | -3.23 [-3.6 to -2.86] | -3.02 [-3.45 to -2.59]
  day 42 results | 4.25 [3.80 to 4.70] | 4.32 [3.84 to 4.79]
Statistical Analysis 1: Comparison: Abbreviated Zagreb (2-1-1) vs Conventional Essen(1-1-1-1-1); Test type: Non-Inferiority or Equivalence — The null hypothesis states that the Zagreb schedule is inferior to the Essen schedule in terms of day 7 antibody titers assuming no difference between the two schedules and the equivalence limit of 1.5 titer levels (log2); ANOVA; ratio of log2 mean (day7) = -0.21, 95% CI 2-sided [-0.77 to 0.35] — Ratio of log2 means (Zagreb/Essen) on day 7
Statistical Analysis 2: Comparison: Abbreviated Zagreb (2-1-1) vs Conventional Essen(1-1-1-1-1); Test type: Non-Inferiority or Equivalence — The null hypothesis states that the Zagreb schedule is inferior to the Essen schedule in terms of day 42 antibody titers assuming no difference between the two schedules and the equivalence limit of 1.5 titer levels (log2); ANOVA; ratio of log2 mean (day 42) = -0.07, 95% CI 2-sided [-0.72 to 0.58] — Ratio of log2 mean (Zagreb/(Essen) on day 42

3. Primary Outcome: Number of Participants Who Reported a Local or Systemic Reaction After Any Vaccination
Description: Specified local and systemic reactions were solicited for 7 days after each vaccination. Number of participants were calculated who reported a local or systemic reaction after any of the vaccinations.
Time Frame: 7 days after each vaccination
Population: Safety was analyzed for the safety set. One enrolled subject was not vaccinated and not included in the safety set because of inappropriate inclusion.
Measure: Number; unit: participants
Arm/Group | Abbreviated Zagreb (2-1-1) | Conventional Essen(1-1-1-1-1)
Number analyzed (Participants) | 549 | 275
participants
  Any local reaction | 483 | 241
  Erythema | 37 | 18
  Swelling | 42 | 38
  Pain | 475 | 236
  Any systemic reaction | 177 | 103
  Chills | 21 | 8
  Malaise | 35 | 17
  Headache | 91 | 49
  Nausea | 28 | 24
  Myalgia | 29 | 23
  Arthralgia | 13 | 13
  Fatigue | 61 | 34
  Rash | 3 | 33
  Fever ≥37.1°C | 124 | 68

4. Secondary Outcome: Percentages of Participants With Seroconversion (Rabies Virus Neutralizing Antibody Concentrations Equal and Above 0.5 IU/ml) on Days 7, 14 and 42.
Description: Percentages of participants with seroconversion (defined as rabies virus neutralizing antibody concentrations equal and above 0.5 IU/ml) on days 7, 14 and 42.
Time Frame: 7 days, 14 days and 42 days
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentages of participants
Arm/Group | Abbreviated Zagreb (2-1-1) | Conventional Essen(1-1-1-1-1)
Number analyzed (Participants) | 69 | 70
percentages of participants
  day 7 | 10.14 [4.18 to 19.79] | 10.0 [4.12 to 19.52]
  day 14 | 100 [94.79 to 100] | 97.14 [90.19 to 99.66]
  day 42 | 100 [94.79 to 100] | 100 [94.87 to 100]

ADVERSE EVENTS:
Time Frame: Any unsolicited adverse events were collected for 7 days after each vaccination, all serious adverse events were collected throughout the whole study period (beyond individual study participation, from 12 Nov 2008 to 12 Jan 2009).
Description: Subjects were instructed to report on a daily basis any adverse events and record them on a diary card.
Arm/Group | Abbreviated Zagreb (2-1-1) | Conventional Essen(1-1-1-1-1)
Serious Adverse Events (participants affected / at risk) | 0/549 | 1/275
Other Adverse Events (participants affected / at risk) | 52/549 | 26/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abbreviated Zagreb (2-1-1) (N=549) | Conventional Essen(1-1-1-1-1) (N=275)
Injury of soft tissue in the leg and shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Safety was analyzed for the safety set. One enrolled subject in the abbreviated Zaghreb group was not vaccinated and not included in the safety set, because of inappropriate inclusion.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abbreviated Zagreb (2-1-1) (N=549) | Conventional Essen(1-1-1-1-1) (N=275)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 52 (52) | 26 (26) — Safety was analyzed for the safety set. One enrolled subject in the abbreviated Zaghreb group was not vaccinated and not included in the safety set, because of inappropriate inclusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less